CLINICAL TRIAL: NCT04555707
Title: The Maintenance Effect of Enstilar Foam in Combination With Otezla
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENS-2001
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Otezla + Enstilar (Experimental)
  Interventions: Drug: Apremilast 30mg; Drug: calcipotriene and betamethasone dipropionate

INTERVENTIONS:
Drug: Apremilast 30mg — 30mg PO BID started within 10 days of baseline
  Other Names: Otezla
Drug: calcipotriene and betamethasone dipropionate — 1 application daily starting at baseline and continuing for 4 weeks; those achieving clear or almost clear PGA at week 4 will continue application twice weekly on Monday and Thursday in combination with Otezla. Enstilar application is discontinued at week 16 and study participation continues until week 20.
  Other Names: Enstilar

SUMMARY:
This is a single-center, open-label study. Approximately 30 qualified subjects will be enrolled in a study lasting 20 weeks which investigates the effect of Enstilar used in combination with Otezla to treat psoriasis.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled in a single-center, open-label study of the treatment of psoriasis. There will be a screening/baseline, week 4, week 16 and week 20 visits. Subjects will include those who have been started on commercial Otezla within the last 10 days of baseline. We will add Enstilar foam QD at baseline visit for 4 weeks. Those subjects who achieve clear or almost clear on PGA scale at week 4 will continue on maintenance dose of Enstilar twice weekly on Mondays and Thursdays QD for the next 12 weeks and they will also continue on Otezla. Subjects will continue to week 20 after stopping Enstilar at week 16..

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female subjects of any race, 18 years of age or higher. Female subjects of childbearing potential must have a (-)UPT result at within 7 days of the first dose of study drug and practice a reliable method of contraception throughout the study;

   A female is considered of childbearing potential unless she is:

   - postmenopausal > 5Y, without a uterus and/or both ovaries; or has been surgically sterile for > 6M.

   Reliable methods of contraception are:

   - hormonal methods or IUD in use > 90d prior to study drug administration, barrier methods plus spermicide in use > 14d prior, or vasectomized partner.

   [Exception: Female subjects of CBP who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counseled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.]
2. Subjects with moderate plaque type psoriasis who have been started on commercial Otezla within the last 10 days
3. Physician Global Assessment (PGA) score of 3
4. Able to understand study requirements and sign Informed Consent/HIPAA forms

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study
2. History of hypercalcemia or Vitamin D toxicity or history of significant renal or hepatic disease
3. Patients with guttate, erythrodermic, or pustular psoriasis
4. Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator.)
5. Skin conditions (e.g. eczema) that may interfere with evaluations of psoriasis
6. Known hypersensitivity to Enstilar Foam or any of its components
7. Current drug or alcohol abuse (Investigator opinion.)
8. Subject unable to commit to all the assessments required by the protocol
9. Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who are clear or almost clear on Physicians Global Assessment at Week 4 | 4 weeks
  Physician assessment of disease severity. 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate

SECONDARY OUTCOMES:
Percent of subjects who are clear or almost clear at week 4, 16 and week 20 on Physicians Global Assessment | week 4, week 16, week 20
  Physician assessment of disease severity. 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate
The percent of subjects who are clear or almost clear at week 4, 16 and week 20 on Patient Global Assessment | week 4, week 16, week 20
  Patient's Global Assessment of Disease Severity. 0=Clear, 1=Very mild, 2=Mild, 3=Moderate, 4=Severe
Percent of subjects who achieve PASI (psoriasis area and severity index) 75 at week 4 | 4 weeks
  The Psoriasis Area and Severity Index (PASI) is a quantitative rating score for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. PASI 75 evaluates if the subject had a 75% or more reduction in their PASI score from baseline.
Percent of subjects who achieve PASI 75 at week 16 | 16 weeks
  The Psoriasis Area and Severity Index (PASI) is a quantitative rating score for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. PASI 75 evaluates if the subject had a 75% or more reduction in their PASI score from baseline.
DLQI (dermatology life quality index) at week 4 | 4 weeks
  The Dermatology Life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored on a four-point Likert scale:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0, Question unanswered = 0. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
DLQI at week 16 | 16 weeks
  The Dermatology Life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored on a four-point Likert scale:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0, Question unanswered = 0. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Itch VAS (visual analogue scale) at week 4 and week 16 | 4 week, 16 weeks
  The VAS is a scale consisting of a 10cm long line and a single question used for measuring itch intensity. The left end point represents "no itch" and the right end point the "worst imaginable itch".

CONTACTS AND LOCATIONS:
Overall Officials: L.H. Kircik, M.D., Principal Investigator — Skin Sciences, PLLC
Locations (1):
- Skin Sciences, PLLC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No